CLINICAL TRIAL: NCT06013813
Title: Adverse Clinical Outcomes Associated With Conventional Versus Distal Radial Access in Patients With Acute Coronary Syndrome With ST-segment Elevation Treated by Percutaneous Coronary Intervention
Brief Title: Conventional vs. Distal Radial Access Outcomes in STEMI Patients Treated by PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Guering Eid Lidt, Director of Cardiac Catheterization Lab, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1367
Record Dates: First submitted 2023-08-08; First posted 2023-08-28 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Myocardial Infarction; Acute Coronary Syndrome
Keywords: STEMI; distal radial access; conventional radial access; MACE
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal radial approach (Experimental): * Clean and dry the puncture site.
  * Simple lidocaine 2% is infiltrated.
  * The artery is punctured in the radial distal zone, and a 6 Fr hydrophilic radial introducer is placed with the Seldinger technique.
  * Verapamil 2.5 mg and Heparin 5000 IU are administered.
  * PCI is performed.
  * Finally, the introducer is withdrawn with the patent hemostasis technique, and a radial compression device is placed (prelude mostly or terumo).
  Interventions: Procedure: Radial Artery approach on percutaneous coronary intervention (PCI)
- Conventional radial approach (proximal radial approach). (Active Comparator): * Clean and dry the puncture site.
  * Simple lidocaine 2% is infiltrated.
  * The artery is punctured in the radial proximal zone, and a 6 Fr hydrophilic radial introducer is placed with the Seldinger technique.
  * Verapamil 2.5 mg and Heparin 5000 IU are administered.
  * PCI is performed.
  * Finally, the introducer is withdrawn with the patent hemostasis technique, and a radial compression device is placed (terumo).
  Interventions: Procedure: Radial Artery approach on percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Radial Artery approach on percutaneous coronary intervention (PCI) — * Randomized patients with a right patent radial artery.
  * The outcomes of the distal radial approach will be compared with those of the conventional radial approach.
  * Technique and devices (introducer and compression devices) are the same in both approaches.

SUMMARY:
This clinical trial aims to compare conventional radial access versus distal radial access in patients with STEMI undergoing PCI. The main question it aims to answer is:

• Mayor adverse cardiac events (MACE) at 30 days in STEMI patients treated by PCI are not inferior when comparing the distal radial approach versus the conventional radial approach ?

Participants will:

* sign the informed consent to enroll in the clinical trial.
* will agree to be treated by PCI
* will be randomized 1:1 to perform PCI by conventional radial or distal radial approach.

If there is a comparison group:

Researchers will compare conventional radial access vs distal radial access to see if the distal approach is not inferior compared to the conventional radial access in order to offer less or equal MACE and a similar rate of a successful procedure.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients underwent PCI.
* Patent radial access (distal and conventional)
* Patients who agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Cardiogenic shock.
* Previous coronary artery bypass grafting (CABG).
* Absence of palpable radial pulse.
* Arteriovenous fistula for hemodialysis.
* Previous radial artery occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2922 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Composite of adverse events of all-cause mortality, myocardial infarction, cerebral vascular event, BARC 3-5 (Bleeding Academic Research Consortium), myocardial infarction and cerebrovascular event, bleeding measure will be with BARC classification. | 24 hours and 30 days after PCI.
  At 24 hours and 30 days after the procedure, patients will be evaluated by radial doppler ultrasonography, lab test, and interrogation of clinical adverse events during hospital stay or 30 days after PCI.

SECONDARY OUTCOMES:
Incidence of myocardial infarction after the procedure | 24 hours to 30 days after PCI
  A new STEMI event is an event that meets the fourth definition of a myocardial infarction according to the current guidelines.
Incidence of cerebral vascular event (hemorrhagic or ischemic stroke) after the procedure | 24 hours to 30 days after PCI.
  Diagnosed by a doctor based on clinical symptoms and imaging tests (CT scan).
Urgent TVR (Revascularization of the treated vessel) | If the patient requires repeat catheterisation for myocardial infarction within the first 30 days after PCI.
  Diagnosed by coronary angiography or intracoronary imaging (IVUS/OCT) showing a complication related to the culprit vessel of the initial event.
Definite stent thrombosis | If the patient requires repeat catheterisation for myocardial infarction within the first 30 days after PCI.
  Diagnosed by coronary angiography or intracoronary imaging (IVUS/OCT) showing a complication related to the culprit vessel of the initial event.
Bleeding assessed by BARC 3-5 to 30 days of evolution in patients with STEMI who received interventional treatment via RD access versus RC access. | 24 hours to 30 days after PCI.
  Evaluated by BARC scale will be used to classify the severity of bleeding into types 0-5 (3-5 are the most important criteria for the clinical trial will define the worse outcome ) Type 0 = no evidence of bleeding Type 1 = minimal bleeding Type 2 = clinically evident bleeding other than 3, 4 or 5 Type 3 = with haematocrit fall ≥ 3g% and/or hemodynamic compromise and/or requiring transfusion and/or intracranial or intraocular bleeding Type 4 = associated with Myocardial Revascularization Surgery Type 5 = fatal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Guering Eid Lidt, PhD, Study Chair — Guering Eid-Lidt
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD will be shared
Supporting Information: Study Protocol, SAP
Time Frame: january 2025 to january 2026
Access Criteria: IPD will be shared for related studies, without distinctions in the nature of each study, information may be freely requested directly by e-mail and each request will be evaluated by the principal investigator of the study.

REFERENCES:
- [Background] Mason PJ, Shah B, Tamis-Holland JE, Bittl JA, Cohen MG, Safirstein J, Drachman DE, Valle JA, Rhodes D, Gilchrist IC; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; and Council on Genomic and Precision Medicine. An Update on Radial Artery Access and Best Practices for Transradial Coronary Angiography and Intervention in Acute Coronary Syndrome: A Scientific Statement From the American Heart Association. Circ Cardiovasc Interv. 2018 Sep;11(9):e000035. doi: 10.1161/HCV.0000000000000035. PMID 30354598
- [Background] Mamas MA, Anderson SG, Carr M, Ratib K, Buchan I, Sirker A, Fraser DG, Hildick-Smith D, de Belder M, Ludman PF, Nolan J; British Cardiovascular Intervention Society; National Institute for Cardiovascular Outcomes Research. Baseline bleeding risk and arterial access site practice in relation to procedural outcomes after percutaneous coronary intervention. J Am Coll Cardiol. 2014 Oct 14;64(15):1554-64. doi: 10.1016/j.jacc.2014.05.075. PMID 25301457
- [Background] Ferrante G, Rao SV, Juni P, Da Costa BR, Reimers B, Condorelli G, Anzuini A, Jolly SS, Bertrand OF, Krucoff MW, Windecker S, Valgimigli M. Radial Versus Femoral Access for Coronary Interventions Across the Entire Spectrum of Patients With Coronary Artery Disease: A Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2016 Jul 25;9(14):1419-34. doi: 10.1016/j.jcin.2016.04.014. Epub 2016 Jun 29. PMID 27372195
- [Background] Valgimigli M, Gagnor A, Calabro P, Frigoli E, Leonardi S, Zaro T, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Cortese B, Sganzerla P, Lupi A, Galli M, Colangelo S, Ierna S, Ausiello A, Presbitero P, Sardella G, Varbella F, Esposito G, Santarelli A, Tresoldi S, Nazzaro M, Zingarelli A, de Cesare N, Rigattieri S, Tosi P, Palmieri C, Brugaletta S, Rao SV, Heg D, Rothenbuhler M, Vranckx P, Juni P; MATRIX Investigators. Radial versus femoral access in patients with acute coronary syndromes undergoing invasive management: a randomised multicentre trial. Lancet. 2015 Jun 20;385(9986):2465-76. doi: 10.1016/S0140-6736(15)60292-6. Epub 2015 Mar 16. PMID 25791214
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Background] Mehta SR, Jolly SS, Cairns J, Niemela K, Rao SV, Cheema AN, Steg PG, Cantor WJ, Dzavik V, Budaj A, Rokoss M, Valentin V, Gao P, Yusuf S; RIVAL Investigators. Effects of radial versus femoral artery access in patients with acute coronary syndromes with or without ST-segment elevation. J Am Coll Cardiol. 2012 Dec 18;60(24):2490-9. doi: 10.1016/j.jacc.2012.07.050. Epub 2012 Oct 24. PMID 23103036
- [Background] Ferrante G, Condello F, Rao SV, Maurina M, Jolly S, Stefanini GG, Reimers B, Condorelli G, Lefevre T, Pancholy SB, Bertrand O, Valgimigli M. Distal vs Conventional Radial Access for Coronary Angiography and/or Intervention: A Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2022 Nov 28;15(22):2297-2311. doi: 10.1016/j.jcin.2022.09.006. PMID 36423974
- [Background] Eid-Lidt G, Rivera Rodriguez A, Jimenez Castellanos J, Farjat Pasos JI, Estrada Lopez KE, Gaspar J. Distal Radial Artery Approach to Prevent Radial Artery Occlusion Trial. JACC Cardiovasc Interv. 2021 Feb 22;14(4):378-385. doi: 10.1016/j.jcin.2020.10.013. PMID 33602433
- [Background] Bernat I, Aminian A, Pancholy S, Mamas M, Gaudino M, Nolan J, Gilchrist IC, Saito S, Hahalis GN, Ziakas A, Louvard Y, Montalescot G, Sgueglia GA, van Leeuwen MAH, Babunashvili AM, Valgimigli M, Rao SV, Bertrand OF; RAO International Group. Best Practices for the Prevention of Radial Artery Occlusion After Transradial Diagnostic Angiography and Intervention: An International Consensus Paper. JACC Cardiovasc Interv. 2019 Nov 25;12(22):2235-2246. doi: 10.1016/j.jcin.2019.07.043. PMID 31753298
- [Background] Eid-Lidt G, Reyes-Carrera J, Farjat-Pasos JI, Saenz AL, Bravo CA, Rangel SN, Salido DZ, Vega Servin NS, Soto-Lopez ME, Gaspar J. Prevention of Radial Artery Occlusion of 3 Hemostatic Methods in Transradial Intervention for Coronary Angiography. JACC Cardiovasc Interv. 2022 May 23;15(10):1022-1029. doi: 10.1016/j.jcin.2022.03.011. PMID 35589232
- [Background] Aminian A, Sgueglia GA, Wiemer M, Kefer J, Gasparini GL, Ruzsa Z, van Leeuwen MAH, Ungureanu C, Leibundgut G, Vandeloo B, Kedev S, Bernat I, Ratib K, Iglesias JF, Al Hage E, Posteraro GA, Pascut D, Maes F, Regazzoli D, Kakonyi K, Meijers TA, Colletti G, Krivoshei L, Lochy S, Zafirovska B, Horak D, Nolan J, Degrauwe S, Tobita K, Saito S. Distal Versus Conventional Radial Access for Coronary Angiography and Intervention: The DISCO RADIAL Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1191-1201. doi: 10.1016/j.jcin.2022.04.032. Epub 2022 May 17. PMID 35595673
- [Result] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Result] Writing Committee Members; Lawton JS, Tamis-Holland JE, Bangalore S, Bates ER, Beckie TM, Bischoff JM, Bittl JA, Cohen MG, DiMaio JM, Don CW, Fremes SE, Gaudino MF, Goldberger ZD, Grant MC, Jaswal JB, Kurlansky PA, Mehran R, Metkus TS Jr, Nnacheta LC, Rao SV, Sellke FW, Sharma G, Yong CM, Zwischenberger BA. 2021 ACC/AHA/SCAI Guideline for Coronary Artery Revascularization: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 Jan 18;79(2):e21-e129. doi: 10.1016/j.jacc.2021.09.006. Epub 2021 Dec 9. PMID 34895950

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT06013813/Prot_SAP_000.pdf